CLINICAL TRIAL: NCT01544777
Title: Visual Quality Following Aspheric and Monovision Lens Implantation - a Comparative Clinical Study
Brief Title: Visual Quality Following Aspheric Intraocular Lens (IOL) Implantation - a Comparative Clinical Study
Acronym: 751
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoya Surgical Optics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: DOF-1
Record Dates: First submitted 2012-02-21; First posted 2012-03-06 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2012-08

CONDITIONS: Aphakia; Cataract
Keywords: Aphakia; Cataract
MeSH Terms: conditions — Aphakia; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Both Eyes (Experimental): Model 751 IOL implanted in both eyes.
  Interventions: Device: Study IOL
- Single eye (Experimental): Model 751 IOL in one eye
  Interventions: Device: Hoya iSert 751
- Control (Active Comparator): Aphakia treatment by negatively aspheric IOL implant, Hoya iSert model 251 or equivalent
  Interventions: Device: Negatively aspheric IOL

INTERVENTIONS:
Device: Study IOL — Aspheric IOL for correction of aphakia
  Other Names: Hoya iSert 751 IOL
  Arms: Both Eyes
Device: Hoya iSert 751 — Model 751 in one eye, standard IOL in other eye
  Other Names: Hoya iSert Model 751
  Arms: Single eye
Device: Negatively aspheric IOL — Negatively aspheric IOL in both eyes
  Other Names: Hoya iSert model 251 or equivalent
  Arms: Control

SUMMARY:
To evaluate visual acuity and quality of vision in participants undergoing cataract surgery with a Hoya model 751 intra-ocular lens and to compare the visual results to the common monofocal lens in use.

ELIGIBILITY:
Inclusion Criteria:

* Senile cataract
* Patient identified as a candidate for cataract surgery and IOL implantation
* Willing to sign informed consent document approved by the Ethical Committee
* Willing to complete all required tests and exams per this protocol

Exclusion Criteria:

* Amblyopia
* History or evidence of any ocular disease that may affect visual acuity
* Previous ocular surgery, including refraction surgery
* Ocular anomalies (e.g. microphthalmos, kerataconous)
* Subjects with greater than 1.0 D of corneal astigmatism
* Subjects who experience intraoperative complications that could affect postoperative IOL centration or tilt

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Uncorrected Visual Acuity (UCVA) (ETDRS)for distance, intermediate and near | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Graham Barrett, MD, Principal Investigator — Sir Charles Gairdner Hospital, Nedlans WA
Locations (1):
- Sir Charles Gairdner Hospital, Nedlands, Western Australia, Australia